CLINICAL TRIAL: NCT02239718
Title: Novel Use of 2-unit Cantilever Resin-bonded Bridges for Replacing Missing Molar Teeth - a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dr Michael G. Botelho, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17100314
Record Dates: First submitted 2014-09-04; First posted 2014-09-15 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Missing Teeth
Keywords: Resin bonded bridges; Clinical trial; Prospective; Survival; Oral health related quality of life
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-unit cantilevered resin bonded bridge (Experimental): Use one tooth as abutment tooth to replace one adjacent missing tooth
  Interventions: Procedure: 2-unit cantilevered resin bonded bridge
- 3-unit fixed movable resin bonded bridge (Active Comparator): Use teeth from both side of the missing tooth space to replace a tooth. The prosthesis is cast in two piece and connected with a fixed-movable joint (semi-precision, allow degree of movement).
  Interventions: Procedure: 3-unit fixed movable resin bonded bridge

INTERVENTIONS:
Procedure: 2-unit cantilevered resin bonded bridge — Use one tooth as abutment tooth to replace one adjacent missing tooth
  Arms: 2-unit cantilevered resin bonded bridge
Procedure: 3-unit fixed movable resin bonded bridge — Use teeth from both side of the missing tooth space to replace a tooth. The prosthesis is cast in two piece and connected with a fixed-movable joint (semi-precision, allow degree of movement).
  Arms: 3-unit fixed movable resin bonded bridge

SUMMARY:
Tooth replacement is a significant issue in the World and while dental implants and conventional bridges have been used to replace missing teeth, dental implants are too expensive for many and conventional dental bridges are destructive to supporting tooth tissue.

Resin-bonded bridges (RBBs) are a conservative and cost effective replacement option that involves minimal tooth preparation, leaving the majority of the tooth intact. They are secured in place with an adhesive cement, which is bonded to the outer enamel layer. Clinical audit of these prostheses at the University of Hong Kong shows two-unit RBBs to have some of the highest success rates in the dental literature for the replacement of missing premolar and incisor teeth. However, for the replacement of molar teeth, two-unit RBBs are not performed, as established protocol and recognised texts contraindicate their use due to concerns with tipping or drifting of supporting teeth. Replacement of a single missing molar tooth can be with a three-unit, fixed-fixed (single-piece casting) or three-unit, fixed-movable (two-part casting). However, the fixed-fixed option has a higher debond failure rate than two-unit RBBs and therefore, at this centre, a modified, 3-unit fixed-movable design is used. This two-part casting allows for minor, independent movements of the supporting teeth and thereby aims to reduce stresses between them and, similarly, reduce de-bonding forces. This has the potential for greater longevity and easier long-term maintenance as if the major part of the bridge debonds it can be recemented.

The aim of this unique study is to compare 2-unit and 3-unit RBBs for the replacement of single missing molar tooth in a randomized clinical trial. These two designs will be clinically evaluated at 6 months , 1 year, 2 years and 3 years to observe the outcome measures. The primary outcome will examine the success of the dental prostheses with respects to the need of any clinical intervention to repair or remediate the RBB or supporting tooth. Minor outcome measures will examine fatigue or damage to the prosthesis, changes in bone support, pulpal or periodontal health or tooth mobility. Patient satisfaction and quality of life evaluation of the dental prostheses will also be examined. Will 2-unit RBBs offer patients a simpler, cheaper, and successful option over current designs? This has not been previously reported.

ELIGIBILITY:
Inclusion Criteria:

1. A missing molar tooth that ranges in length from 8-10 mm as judged by the pre-treatment study model. (No more than one per quadrant, if more than one, then different designs will be used in the same mouth.)
2. The patient has been informed of the various treatment options (dental implants, partial dentures, conventional fixed prosthodontics and no treatment) and if the patient has chosen the RBB as their preferred treatment option, they will be invited to participate in the study
3. The patient is available to attend for clinical examination at 6 monthly interviews for a period up to 36 months from the start of the study
4. The patient will have a minimum of 12 occluding pairs of teeth (24 teeth in total)
5. have a natural dentition opposing the planned RBB
6. More than 30% bone support on the tooth abutment(s)
7. Patients will agree to being randomly assigned to one of the two treatment groups, a 2-unit bridge or 3-unit fixed movable bridge
8. The patient will have been informed on the nature of the study and be required to sign a consent form agreeing to undertake treatment in the study
9. The patient is over 18 years old
10. The patient is in sound dental health, ie no active caries and controlled periodontal disease

Exclusion Criteria:

1. Patients with active tooth decay
2. Patients with uncontrolled periodontal disease. RBB abutment with a probing depth greater than 5mm and bleeding on probing
3. Patients with teeth missing opposite to the planned RBB
4. Abutment tooth mobility of 2 or greater (Millers classification)
5. Patients with a known allergy to the dental alloy used to make the RBB, ie. Ni/Cr
6. Patients with debilitating illnesses or complicating medical conditions
7. Non-vital or root treated abutment teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Survival of bridges (RBB) | Three years
  Clinically whether the bridge is in subject's mouth. Any complication(s) and associated treatment(s) will be recorded. In case where there is absence of complication/treatment, this bridge is regarded as success.
  If complication occur and/or treatment (apart from routine periodontal maintenance) is required but the original bridge is still in the mouth, this bridge is regarded as survival.
  If lost of the original bridge/abutment tooth (teeth) or complication dedicates the remake of the bridge, the bridge is regarded as failed.
  These will be presented in time to fail (survival) as well as time to complication/treatment (success) by Kaplan Meier curves.
Drifting of abutment teeth after insertion of the bridge | Three years
  Models will be taken after insertion/cementation of bridge (RBB) (baseline model) and at review appointments (see Time Frame).
  Vacuum suck down will be made on the baseline model and fitted in subject's mouth during review appointments to screen for any potential tooth movement.
  In potential tooth movement case, models will be scanned and superimposed for analysis of tooth movement (direction and magnitude of movement)

SECONDARY OUTCOMES:
Complications | Three years
  Complications related to the abutment teeth / prosthesis (RBB)
  This is measured from review examinations as well as from patient history (any treatment of the RBB by the third parties other than the study centres)
  Review examination will look for: debonding, fracture of framework, fracture of veneer material, caries occurring related to retainer on the abutments, extraction related to periodontal disease or root fracture resulting in loss of the entire reconstruction, abutment endodontic or apical radiolucency, probing depth greater than 5mm
Abutment mobility | Three years
  Tested by two handles of mirror (Grade 0, I, II, III) and periotest (Grade 0: -8 to +9; I: 10 to 19; II: 20 to 29; III: 30-50)
Proximal contact tightness of the abutments | Three years
  Measured with passing a dental floss and digital tension gauge on metal matrix band
Oral Health related Quality of Life | Three years
  Measured by Oral Health Impact Profile 49 (OHIP) and 14-item satisfaction (Visual Analogue Scale VAS)
  OHIP will involve pre-operative (before treatment) as well as peri-operative (after tooth preparation and before RBB cementation) time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Botelho, BDS MSc PhD, Study Chair — Oral Rehabilitation, Faculty of Dentistry, The University of Hong Kong; Edward CM Lo, BDS MDS PhD, Study Director — Dental Public Health, Faculty of Dentistry, The University of Hong Kong; Yan Wang, BDS MDS PhD, Study Director — Department of Prosthodontics, Guanghua School of Stomatology, Sun Yat-sen University; Walter YH Lam, BDS MDS, Principal Investigator — Oral Rehabilitation, Faculty of Dentistry, The University of Hong Kong
Locations (2):
- China (2):
  - Department of Prosthodontics, Guanghua School of Stomatology & Affiliated Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong
  - Oral Rehabilitation, Faculty of Dentistry, The University of Hong Kong, Hong Kong, Guangdong

REFERENCES:
- [Background] Botelho MG, Ma X, Cheung GJ, Law RK, Tai MT, Lam WY. Long-term clinical evaluation of 211 two-unit cantilevered resin-bonded fixed partial dentures. J Dent. 2014 Jul;42(7):778-84. doi: 10.1016/j.jdent.2014.02.004. Epub 2014 Mar 28. PMID 24685984
- [Background] Lam WY, Botelho MG, McGrath CP. Longevity of implant crowns and 2-unit cantilevered resin-bonded bridges. Clin Oral Implants Res. 2013 Dec;24(12):1369-74. doi: 10.1111/clr.12034. Epub 2012 Oct 2. PMID 23025467
- [Background] Botelho MG, Leung KC, Ng H, Chan K. A retrospective clinical evaluation of two-unit cantilevered resin-bonded fixed partial dentures. J Am Dent Assoc. 2006 Jun;137(6):783-8. doi: 10.14219/jada.archive.2006.0290. PMID 16803807
- [Background] Botelho MG, Dyson JE. Long-span, fixed-movable, resin-bonded fixed partial dentures: a retrospective, preliminary clinical investigation. Int J Prosthodont. 2005 Sep-Oct;18(5):371-6. PMID 16220800
- [Background] Botelho MG. Improved design of long-span resin-bonded fixed partial dentures: three case reports. Quintessence Int. 2003 Mar;34(3):167-71. PMID 12731596
- [Background] Botelho MG. Inhibitory effects on selected oral bacteria of antibacterial agents incorporated in a glass ionomer cement. Caries Res. 2003 Mar-Apr;37(2):108-14. doi: 10.1159/000069019. PMID 12652048
- [Background] Botelho MG, Nor LC, Kwong HW, Kuen BS. Two-unit cantilevered resin-bonded fixed partial dentures--a retrospective, preliminary clinical investigation. Int J Prosthodont. 2000 Jan-Feb;13(1):25-8. PMID 11203604
- [Derived] Botelho MG, Yon MJY, Mak KCK, Lam WYH. A randomised controlled trial of two-unit cantilevered or three-unit fixed-movable resin-bonded fixed partial dentures replacing missing molars. J Dent. 2020 Dec;103:103519. doi: 10.1016/j.jdent.2020.103519. Epub 2020 Nov 2. PMID 33152408